CLINICAL TRIAL: NCT00001926
Title: Connectivity of Occipital and Somatosensory Cortical Areas in Blind Subjects
Brief Title: The Connection Between Areas in the Brain of Blind Patients
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 990031; 99-N-0031
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2003-11

CONDITIONS: Blindness; Brain Mapping; Healthy
Keywords: Plasticity; Magnetic Stimulation; PET; Blind; Braille; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Blindness

INTERVENTIONS:
Drug: O15
Device: Cadwell rTMS

SUMMARY:
The purpose of this study is to test the belief that specific areas of the brain are connected differently in blind patients than patients with sight. In addition, the study will examine the different anatomical connections between brain areas of patients who became blind early in life versus patients who became blind later.

DETAILED DESCRIPTION:
The purpose of this protocol is to test the hypothesis that the anatomical connectivity of occipital and somatosensory areas in early blind subjects differs from that in subjects who became blind later in life and from that in sighted volunteers.

ELIGIBILITY:
INCLUSION CRITERIA:

Subjects with late blindness.

Subjects with early blindness.

Sighted volunteers.

Age between 18 and 65 years.

EXCLUSION CRITERIA:

Subjects with personal or family history of seizures or other neurological or demyelinating disorders.

Pregnant women tested after urine pregnancy test.

Subjects with metal in the cranium except mouth.

Subjects with intracardiac lines and implanted medication pumps.

Subjects with increased intracranial pressure as evaluated by clinical means.

Subjects with cardiac pacemakers.

Intake or neuroleptics.

Subjects with blindness secondary to degenerative CNS diseases.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 45
Dates: Start 1999-04; Study Completion 2003-11

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Cohen LG, Bandinelli S, Findley TW, Hallett M. Motor reorganization after upper limb amputation in man. A study with focal magnetic stimulation. Brain. 1991 Feb;114 ( Pt 1B):615-27. doi: 10.1093/brain/114.1.615. PMID 2004259
- [Background] Fuhr P, Cohen LG, Dang N, Findley TW, Haghighi S, Oro J, Hallett M. Physiological analysis of motor reorganization following lower limb amputation. Electroencephalogr Clin Neurophysiol. 1992 Feb;85(1):53-60. doi: 10.1016/0168-5597(92)90102-h. PMID 1371745
- [Background] Kew JJ, Ridding MC, Rothwell JC, Passingham RE, Leigh PN, Sooriakumaran S, Frackowiak RS, Brooks DJ. Reorganization of cortical blood flow and transcranial magnetic stimulation maps in human subjects after upper limb amputation. J Neurophysiol. 1994 Nov;72(5):2517-24. doi: 10.1152/jn.1994.72.5.2517. PMID 7884476